CLINICAL TRIAL: NCT07164001
Title: Twins With Specific vs. Traditional Fetal Growth Charts (TWiST): A Randomized Controlled Trial
Brief Title: Twins With Specific vs. Traditional Fetal Growth Charts
Acronym: TWiST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Hiba Mustafa, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 27427
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Twin Pregnancy
Keywords: Twin-Specific Growth Chart; Singleton-Based Growth Chart; Fetal Biometry; Small for Gestational Age; Growth Assessment; Perinatal Outcomes; Randomized Controlled Trial; Prenatal Ultrasound; Twin Gestation

STUDY DESIGN:
Intervention Model Description: Participants with twin pregnancies are randomly assigned to either the intervention arm (twin-specific fetal growth chart) or the control arm (singleton-based fetal growth chart). The two groups will be followed in parallel throughout the study period to compare diagnostic accuracy and clinical outcomes. No crossover between arms will occur. Ultrasound measurements and clinical decision-making will adhere to the assigned chart type.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twin-Specific Growth Chart Group (Experimental): Participants in this arm will receive prenatal ultrasound assessments interpreted using a twin-specific growth chart for estimated fetal weight and biometry. Clinical decisions and perinatal risk assessments will be guided based on twin-specific percentiles.
  Interventions: Other: Twin-Specific Growth Chart Interpretation
- Singleton-Based Growth Chart Group (Active Comparator): Participants in this arm will receive prenatal ultrasound assessments interpreted using a singleton-based growth chart for estimated fetal weight and biometry. Clinical decisions and perinatal risk assessments will be based on singleton percentiles, which represent standard practice in many settings.
  Interventions: Other: Singleton-Based Growth Chart Interpretation

INTERVENTIONS:
Other: Twin-Specific Growth Chart Interpretation — Participants in this arm will have their fetal growth assessed using twin-specific growth charts. These charts account for twin gestation norms and may influence clinical decision-making regarding growth restriction and perinatal management. The intervention does not involve any direct physical procedure or device but rather a change in the interpretation framework of routinely collected ultrasound data.
  Other Names: TWiST-Twin Chart
  Arms: Twin-Specific Growth Chart Group
Other: Singleton-Based Growth Chart Interpretation — Participants in this arm will have their fetal growth assessed using singleton-based growth charts. These charts are commonly used in standard practice but may overestimate growth restriction in twin pregnancies. The intervention does not involve any direct physical procedure or device but alters the interpretation framework for standard prenatal ultrasound findings.
  Other Names: TWiST-Singleton Chart
  Arms: Singleton-Based Growth Chart Group

SUMMARY:
This study aims to compare how well two different types of fetal growth charts work in tracking the growth of twins during pregnancy. These charts help doctors decide if a fetus is growing normally. One type is commonly used for all pregnancies, while the other is specially designed for twin pregnancies. The study will enroll pregnant individuals carrying twins. Participants will be randomly assigned to have their care guided by either the traditional chart or the twin-specific chart. Researchers will compare outcomes such as birth weight, timing of delivery, and newborn health. The goal is to find out if using twin-specific charts can improve care and reduce unnecessary interventions.

DETAILED DESCRIPTION:
Twin pregnancies are at increased risk for growth abnormalities and adverse perinatal outcomes. Despite physiological differences in fetal growth patterns between singleton and twin pregnancies, most clinical decisions in the United States still rely on singleton-based fetal growth charts. This randomized controlled trial (RCT) evaluates whether using twin-specific fetal growth charts to guide clinical care results in better perinatal outcomes compared to using standard singleton-based charts.

Participants will be pregnant individuals with twin gestations receiving routine prenatal care at participating clinical sites. Eligible participants will be randomized to one of two groups: (1) management based on singleton growth charts or (2) management based on twin-specific charts. Both charts will be used to assess fetal growth during ultrasound visits, but only the chart assigned to the participant's group will inform clinical decision-making. Data will be collected on outcomes including birth weight, small-for-gestational-age (SGA) classification, gestational age at delivery, NICU admissions, and neonatal morbidity.

The study aims to determine whether using twin-specific fetal growth standards can reduce the overdiagnosis of growth restriction and the associated risks of iatrogenic preterm delivery and unnecessary interventions. Results may support more tailored approaches to growth assessment in twin pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals with a twin pregnancy of at least 18 weeks gestation.
* Willing and able to provide informed consent.
* Planning to deliver at a participating center.

Exclusion Criteria:

* Major fetal anomalies or known aneuploidy.
* Significant maternal medical conditions that might confound study outcomes.
* Inability to comply with study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-01-28 (Estimated)

PRIMARY OUTCOMES:
Rate of Small for Gestational Age (SGA) Diagnosis Based on Ultrasound Biometry | At delivery (up to 42 weeks gestation)
  The primary outcome is the incidence of small for gestational age (SGA) diagnosis among twin pregnancies, as determined by fetal biometry assessed during prenatal ultrasound using either twin-specific or singleton-based growth charts. SGA is defined as an estimated fetal weight below the 10th percentile for gestational age according to the respective chart used in each study arm.

SECONDARY OUTCOMES:
Rate of Neonatal Composite Morbidity | Delivery through neonatal hospital discharge (up to 28 days of life)
  Composite includes one or more of the following: CPAP use >72 hours, intraventricular hemorrhage (IVH), necrotizing enterocolitis (NEC), neonatal hypoglycemia requiring IV therapy, or neonatal death.
Rate of NICU Admission | At delivery
  Percentage of neonates admitted to the Neonatal Intensive Care Unit (NICU) following delivery, as documented in clinical records.
Birthweight Discordance Between Twins | At delivery
  Defined as the percentage difference in birthweight between the two fetuses in each twin pair. Discordance >20% will be considered clinically significant.
Gestational Age at Delivery | At delivery
  Measured in completed weeks of gestation at the time of birth, based on clinical and ultrasound dating.

CONTACTS AND LOCATIONS:
Overall Officials: Hiba Mustafa, MD, Principal Investigator — Indiana University

IPD SHARING:
Plan to Share IPD: Undecided